CLINICAL TRIAL: NCT05652205
Title: A Phase 3, Multicenter, Randomized, Double-blind, Parallel-group, Safety and Efficacy Study of Linaclotide Versus Placebo in Pediatric Subjects, Ages 2 to 5 Years, With Functional Constipation (FC) With a 24-week Open-label Treatment Extension
Brief Title: A Study to Assess Adverse Events and Change in Symptoms With Linaclotide Versus Placebo in Pediatric Subjects, Ages 2 to 5 Years, With Functional Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Ironwood Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M21-572; 2022-501946-31-00 (Other: EU CT)
Record Dates: First submitted 2022-12-02; First posted 2022-12-15 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Functional Constipation (FC); Chronic Idiopathic Constipation (CIC)
Keywords: Functional Constipation (FC); Linaclotide; AGN-182139; Linzess
MeSH Terms: interventions — linaclotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Part 1 Linaclotide (Experimental): Participants will receive linaclotide for 12 weeks.
  Interventions: Drug: Linaclotide
- Part 1 Placebo (Experimental): Participants will receive placebo for 12 weeks.
  Interventions: Drug: Placebo for Linaclotide
- Part 2 Linaclotide (Experimental): Participants who completed study intervention in Part 1 of this study or the Phase 2 Study LIN-MD-67 will receive 24 weeks of linaclotide exposure.
  Interventions: Drug: Linaclotide

INTERVENTIONS:
Drug: Linaclotide — Capsule; oral
  Arms: Part 1 Linaclotide; Part 2 Linaclotide
Drug: Placebo for Linaclotide — Capsule; oral
  Arms: Part 1 Placebo

SUMMARY:
Functional constipation (FC) is a common healthcare problem in children of all ages, potentially due to genetic predisposition, inadequate fiber and fluid intake, and immobility. Currently, there are no pharmacological therapies approved for the treatment of FC. This study will assess adverse events and change in disease activity with linaclotide therapy in participants with FC.

Linaclotide is an approved drug being developed for the treatment of FC in pediatric patients, ages 2 to 5, who meet modified Rome IV criteria for childhood FC. In Part 1 of this study, participants are placed in 1 of 2 groups, called treatment arms. Each group receives a different treatment. There is a 1 in 2 chance that participants will be assigned to placebo. All participants in Part 2 will receive linaclotide. Approximately 116 participants aged 2 to 5 years with FC will be enrolled in this study at around 45 sites worldwide.

Participants will receive daily doses of oral Linaclotide capsules or matching placebo for 12 weeks in Part 1 of the study. In Part 2, the open label long-term safety extension, participants with FC who completed study intervention in Part 1 of Study M21-572 or the Phase 2 Study LIN-MD-67 will receive linaclotide for 24 weeks.

There may be higher treatment burden for participants in this trial compared to their standard of care (due to study procedures). Participants will attend visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver/parent/guardian/legally authorized representative (LAR) is willing and able to comply with procedures required in this protocol, prior to the initiation of any screening or study-specific procedures. In addition, the caregiver/parent/guardian/LAR who will be completing the electronic diary (eDiary) must be able to read and understand the assessments in the eDiary device and undergo training.
* Participant meets modified Rome IV criteria for FC: For at least 1 month before Screening (Visit 1), the participant has had 2 or fewer defecations (with each defecation occurring in the absence of any laxative, suppository, or enema use during the preceding 24 hours) per week. In addition, at least once per week, participant must meet 1 or more of the following:

  * History of retentive posturing or excessive volitional stool retention.
  * History of painful or hard bowel movements (BMs).
  * Presence of a large fecal mass in the rectum.
  * History of large diameter stools.
  * At least 1 episode of fecal incontinence per week after the acquisition of toileting skills, if applicable.

Exclusion Criteria:

* Participant history of:

  * Celiac disease, or positive serological test for celiac disease or the condition is suspected but has not been ruled out by endoscopic biopsy
  * Cystic fibrosis
  * Hypothyroidism that is untreated or treated with thyroid hormone at a dose that has not been stable for at least 3 months prior to Screening (Visit 1)
  * Down's syndrome or any other chromosomal disorder
  * Active anal fissure (i.e., participant reports having streaks of blood on the stool or on toilet paper and/or pain/crying with BM within 2 weeks prior to Screening). (Note: anal fissures that have resolved at least 2 weeks prior to screening would not be exclusionary.) However, if in the investigator's opinion, an anal fissure(s) may be the primary cause of participant's modified Rome IV FC criteria, the participant would not be eligible to participate in the study.
  * Anatomic malformations (e.g., imperforate anus, anal stenosis, anterior displaced anus)
  * Intestinal nerve or muscle disorders (e.g., Hirschprung disease, visceral myopathies, visceral neuropathies)
  * Neuropathic conditions (e.g., spinal cord abnormalities, neurofibromatosis, tethered cord, spinal cord trauma)
  * Lead toxicity, hypercalcemia
  * Inflammatory bowel disease
  * Childhood functional abdominal pain syndrome
  * Poorly treated or poorly controlled psychiatric disorders that might influence his or her ability to participate in the study
  * Lactose intolerance that is associated with symptoms which could confound the assessments in this study
  * History of cancer. (Note: participants with a history of cancer are allowed provided that the malignancy has been in a complete remission before Randomization (Visit 2). A complete remission is defined as the disappearance of all signs of cancer in response to treatment.)
* Has conditions that could interfere with drug absorption including but not limited to short bowel syndrome.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 123 (Actual)
Dates: Start 2022-12-29 (Actual); Primary Completion 2025-09-02 (Actual); Study Completion 2025-09-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the spontaneous bowel movement (SBM) frequency rate (SBMs/week) observed by the primary caregiver during the double-blind study intervention period. | Baseline to Week 12
  An SBM is defined as a BM that occurs in the absence of laxative, enema, or suppository use on the calendar day of the BM or the calendar day before the BM. The caregiver/parent/guardian/legally authorized representative (LAR) will complete the electronic diary (eDiary), providing data for the SBM frequency rate up to the last dose date equivalent to the 12-week SBM frequency rate.
Number of Participants with Adverse Events (AEs) | Up to Approximately 36 Weeks
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation in which a participant is administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Change from baseline in stool consistency observed by the primary caregiver during the double blind study intervention period | Baseline to Week 12
  The caregiver/parent/guardian/legally authorized representative (LAR) will rate and record in an eDiary the consistency of the stool for each BM using the Bristol Stool Form 7-point scale in which 1=Separate hard lumps, like nuts (hard to pass); 2=Sausage-shaped, but lumpy; 3=Like a sausage but with cracks on its surface; 4=Like a sausage or snake, smooth and soft; 5=Soft blobs with clear cut edges (easy to pass); 6=Fluffy pieces with ragged edges, a mushy stool; and 7=Watery, no solid pieces, entirely liquid.
Change from baseline in straining observed by the primary caregiver during the double-blind study intervention period | Baseline to Week 12
  The caregiver/parent/guardian/LAR will rate and record in an eDiary the amount of straining they observe when the child passes the BM.
Change from baseline in proportion of days with fecal incontinence during the double-blind study intervention period (for participants who have acquired toileting skills during daytime and nighttime or acquired toileting skills during daytime only) | Baseline to Week 12
  Each day the caregiver/parent/guardian/LAR will record incidents of fecal incontinence in an eDiary.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (48):
- United States (38):
  - G & L Research, LLC /ID# 250658, Foley, Alabama
  - Velocity Clinical Research - Phoenix /ID# 266280, Phoenix, Arizona
  - HealthStar Research of Hot Springs PLLC /ID# 249481, Hot Springs, Arkansas
  - Applied Research Center of Arkansas /ID# 249764, Little Rock, Arkansas
  - Advanced Research Center /ID# 249412, Anaheim, California
  - Kindred Medical Institute - Corona /ID# 249485, Corona, California
  - Medical Ctr for Clin Research /ID# 254386, San Diego, California
  - Prohealth Research Center /ID# 249420, Doral, Florida
  - KIDZ Medical Services - Hollywood /ID# 250823, Hollywood, Florida
  - Nemours Children's Health System /ID# 250881, Jacksonville, Florida
  - Kissimmee Clinical Research /ID# 252206, Kissimmee, Florida
  - South Miami Medical & Research Group Inc. /ID# 249418, Miami, Florida
  - Valencia Medical & Research Center /ID# 250452, Miami, Florida
  - Palmetto Professional Research /ID# 250875, Miami, Florida
  - South Florida Research Ph I-IV /ID# 252350, Miami Springs, Florida
  - Velocity Clinical Research Macon /ID# 266516, Macon, Georgia
  - Rophe Adult & Pediatric Medicine /ID# 250663, Union City, Georgia
  - Michael W. Simon, MD, PSC /ID# 250664, Lexington, Kentucky
  - Velocity Clinical Research - Lafayette /ID# 266751, Lafayette, Louisiana
  - Frederick County Pediatrics /ID# 249483, New Market, Maryland
  - Michigan Center of Medical Research /ID# 251088, Farmington Hills, Michigan
  - MNGI Digestive Health, P. A. /ID# 249676, Minneapolis, Minnesota
  - Velocity Clinical Research- Hastings Nebraska /ID# 252132, Hastings, Nebraska
  - Rutgers New Jersey Medical School Campus, Doctors Office Center /ID# 250876, Newark, New Jersey
  - Univ NC Chapel Hill /ID# 252044, Chapel Hill, North Carolina
  - UH Cleveland Medical Center /ID# 250893, Cleveland, Ohio
  - IPS Research Company /ID# 250822, Oklahoma City, Oklahoma
  - Frontier Clinical Research, LLC - Scottdale /ID# 250656, Scottdale, Pennsylvania
  - Frontier Clinical Research - Smithfield /ID# 250657, Smithfield, Pennsylvania
  - Coastal Pediatric Research - West Ashley B /ID# 249413, Charleston, South Carolina
  - Tribe Clinical Research LLC /ID# 255656, Greenville, South Carolina
  - Coastal Pediatric Research - Summerville /ID# 249423, Summerville, South Carolina
  - Tullahoma Pediatrics /ID# 250892, Tullahoma, Tennessee
  - Houston Clinical Research Associates /ID# 250779, Houston, Texas
  - Prime Clinical Research - Mansfield - East Broad Street /ID# 266236, Mansfield, Texas
  - ClinPoint Trials /ID# 250448, Waxahachie, Texas
  - Carilion Medical Center /ID# 249790, Roanoke, Virginia
  - Frontier Clinical Research - Kingwood /ID# 251154, Kingwood, West Virginia
- Bulgaria (5):
  - University Hospital Plovdiv /ID# 250814, Tsentar, Plovdiv
  - UMHAT Kanev /ID# 250815, Rousse
  - Acibadem City Clinic Tokuda University Hospital EAD /ID# 251234, Sofia
  - Specialized Hospital For Active Treatment Of Children Diseases Prof. Ivan Mitev /ID# 251233, Sofia
  - Nova Clinic /ID# 250816, Varna
- Netherlands (2):
  - Amphia Ziekenhuis /ID# 251698, Breda, North Brabant
  - Amsterdam UMC, locatie AMC /ID# 251295, Amsterdam, North Holland
- United Kingdom (3):
  - Disc_Barts Health NHS Trust - The Royal London Hospital /ID# 251179, London, Greater London
  - Doncaster Royal Infirmary /ID# 252080, Armthorpe Road
  - Northern Licolnshire and Goole NHS Foundation Trust /ID# 252007, Grimsby

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — https://www.abbvieclinicaltrials.com/study/?id=M21-572